CLINICAL TRIAL: NCT04036058
Title: Effect of Expanding Barrier Precautions for Reducing Clostridium Difficile Acquisition in VA
Brief Title: Effect of Expanding (Gloving) Barrier Precautions for Reducing Clostridium Difficile Acquisition (and Infection) in VA
Acronym: GLORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 18-087
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; Barrier Precautions; Personal Protective Equipment

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment: the 10 participating units will be randomized; at each site, one unit will be randomized to the intervention group and one unit to the control group so that 5 units will enact the universal gloving intervention and 5 units will continue standard of care gloving practices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Enact universal gloving practices
  Interventions: Other: Universal gloving
- Control (No Intervention): Continue standard of care gloving practices

INTERVENTIONS:
Other: Universal gloving — The intervention will consist of all healthcare workers (nurses, providers, respiratory therapists, radiology and laboratory technicians, etc) utilizing universal gloving (non-sterile gloves) for all patient contacts in the units that are randomized to receive the intervention. If a patient in the intervention unit is known to have CDI or a multidrug-resistant organisms, both gowns and gloves will be used as is currently recommended. Signage denoting what type of precautions are needed will be utilized.
  Other Names: Expanded barrier precautions
  Arms: Intervention

SUMMARY:
Clostridium difficile (C. difficile) is a major pathogen causing serious healthcare-associated diarrheal illness in patients. Prevention of healthcare facility-onset C. difficile infection (CDI) is essential. Many CDI cases are caused by the transmission of the pathogen from patients who carry the bacteria, but do not have symptoms. However, there are limited data on how to prevent the transmission of C. difficile from patients who do not have symptoms. Universal gloving practices - the use of gloves by all healthcare workers for all patient contacts - may reduce CDI cases. In this study, the investigators will examine the effectiveness of universal gloving practices as compared to standard of care (use of gloving for contact only in patients with known CDI or other infections). The investigators will compare the effects of these practices on the transmission of C. difficile within participating hospital units to determine if universal gloving is an effective practice to prevent healthcare-associated CDI.

DETAILED DESCRIPTION:
Background: Clostridium difficile infection (CDI) has become the most common healthcare-associated infection (HAI) in US hospitals, causing approximately 500,000 infections and 30,000 deaths per year. Prevention of healthcare-onset (HO) CDI has quickly become a priority for many hospitals. Hospital prevention measures are limited to modifiable risk factors (i.e., prudent antibiotic use and limiting exposure to C. difficile). Hospital exposure to C. difficile can occur directly (i.e., hands or clothing of healthcare workers) or indirectly (i.e., environmental surfaces or shared equipment), so infection prevention measures focus on healthcare worker hand hygiene, barrier precautions (use of gowns and gloves) and cleaning of the hospital environment and reusable medical equipment. However, these interventions are limited to symptomatic patients who test positive for CDI. Asymptomatic patients serve as a reservoir for cross-contamination, but microbiological screening for asymptomatic carriage of C. difficile is not routinely performed in healthcare. Gloving for all patient contacts may interrupt transmission from asymptomatic patients colonized with C. difficile.

Objectives: The overall purpose of the study is to determine the effectiveness of healthcare worker use of gloves for all patient contact (universal gloving) on reducing acquisition of C. difficile and hospital-onset CDI in inpatient hospital units. The main objective of the study is to compare the effects of universal gloving for all patient contact to the current standard of care (i.e., glove and gown use only for known CDI cases). The specific aims are: 1) compare the effects of universal gloving for all patient contact to the current standard of care on C. difficile acquisition rates in hospitalized patients; 2) compare the effects of universal gloving compared to standard of care on CDI rates, other HAI rates, 30-day mortality, and unit length of stay; and 3) evaluate intervention fidelity, cost, and stakeholder experiences with universal gloving.

Methods: The study will be a cluster randomized trial (CRT) in ten inpatient VA hospital units. Hospital units will be randomized either to implement universal gloving intervention or to continue standard of care. The universal gloving intervention will consist of all healthcare workers (nurses, providers, respiratory therapists, radiology and laboratory technicians, etc) utilizing gloves for all patient contacts in the units that are randomized to receive the intervention. The non-intervention units will follow standard of care which consists of healthcare workers using gowns and gloves only for patients with known CDI and other infections (e.g., MRSA). Unit-level data will be collected, including C. difficile acquisition and infection rates, mortality, length of stay, barrier precaution compliance, and end-user perceptions.

ELIGIBILITY:
Inclusion Criteria:

VA inpatient units meeting the following criteria are eligible to participate in the study:

* Ability to identify one of the following inpatient units as defined by Centers for Disease Control (CDC) National Healthcare Safety Network30 by reviewing prior 12-month patient mix data (at least 80% of patients meet patient type):

  * Adult Acute Medical Ward: Hospital area for the evaluation and treatment of patients with medical conditions or disorders.
  * Adult Acute Medical/Surgical Ward: Hospital area for the evaluation of patients with medical and/or surgical conditions.
  * Adult Acute Surgical Ward: Hospital area for evaluation and treatment of patients who have undergone a surgical procedure.
* Ability to collect and upload data (HAIs, mortality, length of stay, hand hygiene and barrier precaution compliance; glove use and glove plus gown use for contact precautions) required for analysis.
* Local R&D Committee approval.
* Letter of support from the Hospital Director or Chief of Staff.
* Ability to enroll one unit to intervention and one unit to control.

To participate in interviews or focus groups, the individual must be:

* 18 years of age or older
* A patient admitted to the participating unit OR a healthcare worker who has regular work duties on the participating unit.

Exclusion Criteria:

* Intensive care units
* Long term care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (6):
- United States (6):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: inpatient hospital units
Period: Overall Study
Arm/Group | Intervention | Control
Started | 470; 5 inpatient hospital units | 310; 5 inpatient hospital units
Completed | 303; 5 inpatient hospital units | 171; 5 inpatient hospital units
Not Completed | 167; 0 inpatient hospital units | 139; 0 inpatient hospital units

BASELINE CHARACTERISTICS:
Population: participants that are reported in the Participant Flow differ from the baseline analysis population due to missing demographic data
Units Other Than Participants: inpatient hospital units
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 450 | 298 | 748
Number analyzed (inpatient hospital units) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 70 [29 to 100] | 72 [30 to 101] | 71 [29 to 101]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 15 | 58
  Male | 407 | 283 | 690
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 131 | 91 | 222
  White | 278 | 185 | 463
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 31 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: C. Difficile Acquisition Rates
Description: Acquisition will be defined as a patient who has an initial stool culture upon unit admission that is negative for C. difficile and the patient's subsequent discharge culture within the same unit that is positive for C. difficile. Acquisition rate will be (# of acquisitions/patient days)
Time Frame: during hospitalization, approximately 5 days
Population: The intervention group had 5569 patient admissions in 5 participating units with 988 patient days of care; 303 subjects had both admission and discharge specimens with 13 that acquired c. difficile (c. difficile negative upon admission and positive upon discharge). The control group had 4412 patient admissions in 5 participating units with 674 patient days of care; 171 subjects had both admission and discharge specimens with 7 that acquired c. difficile.
Measure: Mean (95% Confidence Interval); unit: C. diff acquisition per patient days
Units Other Than Participants: patient days of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 303 | 171
Number analyzed (patient days of care) | 988 | 674
C. diff acquisition per patient days | 13.2 [6.1 to 20.3] | 10.4 [2.7 to 18.0]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.611, t-test, 2 sided

2. Secondary Outcome: Hospital-onset C. Difficile Infection (HO-CDI) Rates
Description: The development of CDI as determined by the presence of clinical symptoms and positive laboratory results. Infection rates will be measured on the unit level. Infection rate will be (# of CDI/patient days)
Time Frame: monthly, up to 18 months
Population: In the intervention group there were 5369 patient admitted in the 5 participating inpatient hospital units with 37842 patient days of care. The intervention group had 5569 patient admissions in 5 participating units with 37842 patient days of care; 9 subjects developed CDI. The control group had 4412 patient admissions in 5 participating units with 40310 patient days of care; 21 subjects developed CDI.
Measure: Mean (95% Confidence Interval); unit: CDI per patient days
Units Other Than Participants: patient days of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5369 | 4412
Number analyzed (patient days of care) | 37842 | 40310
CDI per patient days | 0.2379 [0.0825 to 0.3932] | 0.5210 [0.2982 to 0.7437]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.0435, t-test, 2 sided

3. Secondary Outcome: MRSA (HAI) Rates
Description: The rates of healthcare-associated methicillin-resistant Staphylococcus aureus (MRSA) infection will be measured as (# of MRSA cases/patient days) on the unit level.
Time Frame: monthly, up to 18 months
Population: The control had 4412 admissions in 5 units with 40310 patient days; 7 subjects developed MRSA.
  The intervention group had 5369 patient admissions in 5 participating units with 37843 patient days of care; 2 subjects developed MRSA. The control group had 4412 patient admissions in 5 participating units with 40310 patient days of care; 7 subjects developed MRSA.
Measure: Mean (95% Confidence Interval); unit: MRSA per patient days
Units Other Than Participants: patient days of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5369 | 4412
Number analyzed (patient days of care) | 37843 | 40310
MRSA per patient days | 0.0528 [-0.0204 to 0.1261] | 0.1737 [0.0450 to 0.3022]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.1158, t-test, 2 sided

4. Secondary Outcome: CLABSI (HAI) Rates
Description: The rates of healthcare-associated central line-associated bloodstream infection (CLABSI) will be measured as (# of CLABSI cases per number of device days) on the unit level.
Time Frame: monthly, up to 18 months
Population: The intervention group had 5569 patient admissions in 5 participating units with 4846 line days of care; 5 subjects developed CLABSI. The control group had 4412 patient admissions in 5 participating units with 5100 line days of care; 1 subjects developed CLABSI.
Measure: Mean (95% Confidence Interval); unit: CLABSI per central line days
Units Other Than Participants: line days of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5569 | 4412
Number analyzed (line days of care) | 4846 | 5100
CLABSI per central line days | 1.0318 [0.1279 to 1.9357] | 0.1961 [-0.1882 to 0.5804]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.0898, t-test, 2 sided

5. Secondary Outcome: CAUTI (HAI) Rates
Description: The rates of healthcare-associated catheter-associated urinary tract infection (CAUTI) will be measured as (# of CAUTI cases per number of device days) on the unit level.
Time Frame: monthly, up to 18 months
Population: The intervention group had 5569 patient admissions in 5 participating units with 4807 catheter days of care; 0 subjects developed CAUTI. The control group had 4412 patient admissions in 5 participating units with 5763 catheter days of care; 3 subjects developed CAUTI.
Measure: Mean (95% Confidence Interval); unit: CAUTI per foley catheter days
Units Other Than Participants: catheter days of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5569 | 4412
Number analyzed (catheter days of care) | 4807 | 5763
CAUTI per foley catheter days | 0.00 [0.0 to 0.0] | 0.5206 [-0.0684 to 1.1095]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.114, t-test, 2 sided

6. Secondary Outcome: Intervention Fidelity - Barrier Precaution Compliance
Description: Healthcare worker barrier precaution compliance with unit-wide gloving practices during patient care activities will be measured via observations in participating units. Compliance will be measured as a percentage of use of appropriate gloving practices per opportunities for gloving practices.
Time Frame: monthly, up to 18 months
Population: This population represents healthcare worker glove compliance (intervention fidelity) rather than patient participant data.
Measure: Mean (95% Confidence Interval); unit: glove compliance per glove observations
Units Other Than Participants: inpatient hospital units
Arm/Group | Intervention
Number analyzed (Participants) | 717
Number analyzed (inpatient hospital units) | 5
glove compliance per glove observations | 0.651 [0.616 to 0.686]

7. Secondary Outcome: 30-day Mortality
Description: Mortality will be defined as the number of patients who die per the number of patient days at risk during study period. Mortality rate will be (# of deaths/patient days)
Time Frame: during hospitalization, up to one month
Population: participants that are reported in the Participant Flow differ from the baseline analysis population due to missing mortality data
Measure: Mean (95% Confidence Interval); unit: patient deaths per patient admission
Units Other Than Participants: inpatient hospital units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 988 | 674
Number analyzed (inpatient hospital units) | 5 | 5
patient deaths per patient admission | 28.3 [18.0 to 38.7] | 38.6 [24.0 to 53.1]

8. Secondary Outcome: Length of Stay
Description: the average number of days spent in the participating unit based on unit admission and unit discharge dates
Time Frame: during hospitalization, approximately 5 days
Measure: Mean (Standard Error); unit: days
Units Other Than Participants: inpatient hospital units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 470 | 310
Number analyzed (inpatient hospital units) | 5 | 5
days | 3.2 (0.295) | 3.6 (0.770)

9. Secondary Outcome: HAI Costs
Description: total costs in U.S. dollars attributed to the number of HAIs during study period
Time Frame: through study completion, an average of 18 months
Population: Overall Number of Participants Analyzed is inconsistent with the total number of participants reported in the Participant Flow module because we used unit-level aggregate data rather than participant-level data.
Measure: Number; unit: U.S. dollars
Units Other Than Participants: inpatient hospital units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5369 | 4412
Number analyzed (inpatient hospital units) | 5 | 5
U.S. dollars | 155349 | 362460

10. Secondary Outcome: Supply Costs
Description: total costs in U.S. dollars attributed to the number of gloves used during study period
Time Frame: through study completion, an average of 18 months
Population: as for outcome 9
Measure: Number; unit: U.S. dollars
Units Other Than Participants: inpatient hospital units
Arm/Group | Intervention
Number analyzed (Participants) | 5369
Number analyzed (inpatient hospital units) | 5
U.S. dollars | 42883

11. Secondary Outcome: Patient and Healthcare Worker Experience
Description: Qualitative data describing the patient and healthcare worker experience with the intervention of universal gloving.
Time Frame: months 12 - 18
Population: there were 15 patient interviews and 23 employee interviews but thematic quantitative analysis was not conducted for employee interviews.
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 15
participants
  patient perceived no change in care | 10
  patient perceived no change in hcw hand hygiene | 10
  patient perceived no change in hcw work activities | 10

ADVERSE EVENTS:
Time Frame: during hospitalization, up to one month
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 28/470 | 26/310
Serious Adverse Events (participants affected / at risk) | 0/470 | 0/310
Other Adverse Events (participants affected / at risk) | 0/470 | 0/310

LIMITATIONS AND CAVEATS:
Central institutional review board (CIRB) determination for written informed consent led to low enrollment numbers; limited 24/7 availability of research coordinators and burden to busy clinicians and hospitalized patients. Therefore, the primary aim (C. difficile acquisition) was not adequately powered to detect differences. Other real-world challenges to study enrollment was the ongoing corona virus disease of 2019 (COVID-19) pandemic which wasn't officially declared over until May 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT04036058/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04036058/ICF_002.pdf